CLINICAL TRIAL: NCT02604459
Title: Does Optimized General Anesthesia Care Reduce Postoperative Delirium In Older Patients Undergoing Hip Fracture Repair?
Brief Title: Does Optimized General Anesthesia Care Reduce Postoperative Delirium?
Acronym: OPCare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited availability of subjects meeting inclusion criteria resulting in early termination (lack of funding) before meeting target enrollment.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Quinn Johnson, Chair, Anesthesiology, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1212915
Record Dates: First submitted 2015-11-04; First posted 2015-11-13 (Estimated); Results first posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Hip Fractures; Anesthesia; Delirium
MeSH Terms: conditions — Hip Fractures; Delirium | interventions — Anesthesia, General; Propofol; Fentanyl; Sevoflurane

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The individuals assessing the patients for delirium after surgery will be unaware of the treatment in the operating room.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Usual general anesthesia care (Active Comparator): Subjects will have their general anesthetic management directed at the discretion of the anesthesia provider.
  General anesthesia with be maintained with propofol, fentanyl, sevoflurane
  Interventions: Procedure: General anesthesia; Drug: propofol; Drug: fentanyl; Drug: sevoflurane
- Optimized general anesthesia care (Experimental): The subjects will have general anesthesia with propofol, fentanyl, sevoflurane. In addition the subjects will be monitored with a depth of anesthesia monitor (BIS) and a cerebral oximeter (Foresight). These additional monitors will be used to direct care. BP management: Systolic BP will be maintained within 20% of baseline systolic BP variables.
  Interventions: Device: cerebral oximeter (Fore-Sight); Device: depth of anesthesia monitor (BIS); Procedure: BP management; Procedure: General anesthesia; Drug: propofol; Drug: fentanyl; Drug: sevoflurane
- Mini Mental State Exam (Active Comparator): Subjects will have their general anesthetic management directed at the discretion of the anesthesia provider.
  General anesthesia with be maintained with propofol, fentanyl, sevoflurane
  Interventions: Procedure: General anesthesia; Drug: propofol; Drug: fentanyl; Drug: sevoflurane
- Tested and Excluded (Other): Subjects will have their general anesthetic management directed at the discretion of the anesthesia provider.
  General anesthesia with be maintained with propofol, fentanyl, sevoflurane
  Interventions: Procedure: General anesthesia; Drug: propofol; Drug: fentanyl; Drug: sevoflurane

INTERVENTIONS:
Device: cerebral oximeter (Fore-Sight) — The cerebral oximeter will be monitored in the optimized care group and cerebral oxygenation will be maintained at 60% or higher.
  Arms: Optimized general anesthesia care
Device: depth of anesthesia monitor (BIS) — The depth of anesthesia will be maintained between 40 and 60 in the optimized care group.
  Arms: Optimized general anesthesia care
Procedure: BP management — The systolic blood pressure will be maintained within 20% of preoperative levels in the optimized care group.
  Arms: Optimized general anesthesia care
Procedure: General anesthesia — General anesthesia will be used in both groups
Drug: propofol — propofol per protocol
  Other Names: diprivan
Drug: fentanyl — fentanyl per protocol
  Other Names: sublimaze
Drug: sevoflurane — maintenance of anesthesia with inhaled sevoflurane
  Other Names: ultane

SUMMARY:
Postoperative delirium occurs in up to 65% of elders undergoing surgery for repair of a hip fracture and this complication is independently associated with increased morbidity, mortality, length of hospital stay, and placement in long-term care institutions. To date, the only intervention shown to be effective at minimizing postoperative delirium is a proactive geriatric consultation. This prospective randomized clinical trial will randomize 160 adults, aged 65 years or older, to either optimized general anesthesia or usual general anesthesia care for hip fracture surgery to determine if the optimized anesthesia management reduces the severity of postoperative delirium.

DETAILED DESCRIPTION:
Subjects will be randomized to one of two intraoperative anesthesia treatment groups: 1.) Usual care - the anesthetic management will be at the discretion of the anesthesia provider; or 1.) Optimal care - the intraoperative depth of anesthesia will be directed using a BIS monitor, blood pressure will be maintained within 20% of preoperative levels, and cerebral oxygenation will be maintained > 60% during anesthesia. Subjects will be evaluated using the Confusion Assessment Method (CAM) for the first 5 postoperative days to determine if they experience postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legal representative has voluntarily signed the informed consent approved by the Institutional Review Board,
* Hip fracture surgery scheduled under general anesthesia
* Subject is 65 years or older on the day of surgery

Exclusion Criteria:

* Inability to follow directions or comprehend the English language
* Severe uncorrected visual or auditory handicaps
* Delirium at screening or baseline
* Emergency surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quinn L Johnson, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospitals, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual General Anesthesia Care: Subjects will have their general anesthetic management directed at the discretion of the anesthesia provider.
  General anesthesia with be maintained with propofol, fentanyl, sevoflurane
  General anesthesia: General anesthesia will be used in both groups
  propofol: propofol per protocol
  fentanyl: fentanyl per protocol
  sevoflurane: maintenance of anesthesia with inhaled sevoflurane
- Mini-Mental State Examination: If a patient is enrolled in the study, but scores < 15 on the MMSE, they will remain in the study but will not be randomized to one of the treatment groups. They will receive the same type of general anesthesia for their hip fracture surgery as that done for randomized subjects. They will not be monitored with bispectral index or cerebral oximetry during the surgical procedure.
Period: Overall Study
Arm/Group | Usual General Anesthesia Care | Optimized General Anesthesia Care | Mini-Mental State Examination | Tested and Excluded
Started | 56 | 53 | 22 | 14
Completed | 56 | 53 | 22 | 14
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis of active comparator arm (usual general anesthesia care) and experimental arm (optimized general anesthesia care).
Groups:
- Active Comparator: Usual General Anesthesia Care; Mini Mental State Exam; Tested and Excluded: Subjects will have their general anesthetic management directed at the discretion of the anesthesia provider.
  General anesthesia with be maintained with propofol, fentanyl, sevoflurane
- Experimental: Optimized General Anesthesia Care: The subjects will have general anesthesia with propofol, fentanyl, sevoflurane. In addition the subjects will be monitored with a depth of anesthesia monitor (BIS) and a cerebral oximeter (Foresight). These additional monitors will be used to direct care. BP management: Systolic BP will be maintained within 20% of baseline systolic BP variables.
- Total: Total of all reporting groups
Arm/Group | Active Comparator: Usual General Anesthesia Care | Experimental: Optimized General Anesthesia Care | Mini Mental State Exam | Tested and Excluded | Total
Number analyzed (Participants) | 56 | 53 | 22 | 14 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.1 (8.4) | 77.8 (9.3) | 86.6 (6.8) | 81 (7.9) | 78 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 36 | 17 | 9 | 105
  Male | 13 | 17 | 5 | 5 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 55 | 53 | 21 | 13 | 142
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
American Society of Anesthesiologists (ASA) Physical Status Classification System [Count of Participants; unit: Participants] — The ASA Physical Status Classification System is used to assess and communicate a patient's pre-anesthesia medical co-morbidities. Scale: 1-6.
  A higher ASA Physical Status score indicates more severe systemic disease. Patients with a higher score is generally at higher risk for complications.
  Participants
    2 | 8 | 10 | 1 | 6 | 25
    3 | 39 | 33 | 16 | 6 | 94
    4 | 9 | 10 | 4 | 1 | 24
    5 | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Severity of Postoperative Delirium
Description: Delirium Rating Scale-Revised-98 (DRS-R-98) is a 16-item clinician-rated scale with 13 severity items and 3 diagnostic items (maximum severity score of 39 points). Higher scores indicate more severe delirium; score of 0 indicates no delirium. Only the number of patients who had high scores on the DRS-R-98 are reported.
Time Frame: 5 postoperative days
Population: Number of patients who presented with postoperative delirium and had high scores on the delirium test measures per group are indicated here. Patients who were excluded were not assessed for postoperative delirium.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Comparator: Usual General Anesthesia Care | Experimental: Optimized General Anesthesia Care | Mini Mental State Exam | Tested and Excluded
Number analyzed (Participants) | 8 | 4 | 14 | 0
score on a scale | 0.14 (0.35) | 0.06 (0.23) | 0.63 (0.49) |

2. Secondary Outcome: Number of Patients Who Presented With Postoperative Delirium
Description: Confusion Assessment Method (CAM) with delirium scored as 'present' (1) or 'absent' (0) based on question responses; CAM is considered positive based on the CAM algorithm: presence of acute onset or fluctuating course, inattention, and disorganized thinking or altered level of consciousness.
Time Frame: 5 postoperative days
Population: Number of patients who presented with postoperative delirium are reported. The patients who where tested and then excluded were not included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Usual General Anesthesia Care | Experimental: Optimized General Anesthesia Care | Mini Mental State Exam | Tested and Excluded
Number analyzed (Participants) | 56 | 53 | 22 | 0
Participants | 8 | 4 | 0 |

3. Secondary Outcome: Perioperative Inflammatory Response
Description: Blood will be drawn for analysis of inflammatory markers including interleukin 6 (IL6), interleukin 10 (IL10), tumor necrosis factor (TNF) alpha on the day prior to surgery, at the end of surgery and on the second postoperative day.
Time Frame: preoperative, day of surgery, and postoperative day 2
Population: Lack of funding prevented the analysis of blood to obtain inflammatory markers.
Arm/Group | Active Comparator: Usual General Anesthesia Care | Experimental: Optimized General Anesthesia Care | Mini Mental State Exam | Tested and Excluded
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Patients Who Experienced Postoperative Complications
Description: The investigators will make a telephone call to the subjects at 3 months and 1 year after surgery to determine if the subject has experienced any complications. We will ask the subjects about the occurrence of infections, strokes, cardiac problems, or respiratory problems since discharge from the hospital.
Time Frame: 3 months and 1 year
Population: Number analyzed in rows differs due to loss to follow-up. Patients who were excluded from the study were not followed op post operatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Comparator: Usual General Anesthesia Care | Experimental: Optimized General Anesthesia Care | Mini Mental State Exam | Tested and Excluded
Number analyzed (Participants) | 56 | 53 | 22 | 0
Participants
  3 Months: Cardiac arrest requiring cardiopulmonary resuscitation: number analyzed (Participants) | 55 | 53 | 19 | 0
  3 Months: Cardiac arrest requiring cardiopulmonary resuscitation | 1 | 0 | 0 |
  3 Months: Myocardial infarction: number analyzed (Participants) | 56 | 53 | 19 | 0
  3 Months: Myocardial infarction | 1 | 1 | 1 |
  3 Months: Both cardiac arrest requiring cardiopulmonary resuscitation and myocardial infarction: number analyzed (Participants) | 56 | 53 | 19 | 0
  3 Months: Both cardiac arrest requiring cardiopulmonary resuscitation and myocardial infarction | 0 | 0 | 0 |
  3 Months: Deep incisional surgical site infection: number analyzed (Participants) | 56 | 53 | 19 | 0
  3 Months: Deep incisional surgical site infection | 0 | 1 | 0 |
  3 Months: Organ/space surgical site infection: number analyzed (Participants) | 56 | 53 | 19 | 0
  3 Months: Organ/space surgical site infection | 1 | 2 | 0 |
  1 Year: Cardiac arrest requiring cardiopulmonary resuscitation: number analyzed (Participants) | 49 | 46 | 16 | 0
  1 Year: Cardiac arrest requiring cardiopulmonary resuscitation | 2 | 0 | 2 |
  1 Year: Myocardial infarction: number analyzed (Participants) | 49 | 46 | 16 | 0
  1 Year: Myocardial infarction | 0 | 1 | 0 |
  1 Year: Both cardiac arrest requiring cardiopulmonary resuscitation and myocardial infarction: number analyzed (Participants) | 49 | 46 | 16 | 0
  1 Year: Both cardiac arrest requiring cardiopulmonary resuscitation and myocardial infarction | 1 | 0 | 0 |
  1 Year: Deep incisional surgical site infection: number analyzed (Participants) | 49 | 46 | 16 | 0
  1 Year: Deep incisional surgical site infection | 1 | 1 | 0 |
  1 Year: Organ/space surgical site infection: number analyzed (Participants) | 49 | 46 | 16 | 0
  1 Year: Organ/space surgical site infection | 0 | 2 | 0 |

ADVERSE EVENTS:
Time Frame: 1 year
Description: Patients who were excluded from the study were not followed up for adverse events or all-cause mortality.
Arm/Group | Active Comparator: Usual General Anesthesia Care | Experimental: Optimized General Anesthesia Care | Mini Mental State Exam | Tested and Excluded
All-Cause Mortality (participants affected / at risk) | 8/56 | 6/53 | 10/22 | 0/0
Serious Adverse Events (participants affected / at risk) | 26/56 | 28/53 | 11/22 | 0/0
Other Adverse Events (participants affected / at risk) | 25/56 | 20/53 | 0/22 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Usual General Anesthesia Care (N=56) | Experimental: Optimized General Anesthesia Care (N=53) | Mini Mental State Exam (N=22) | Tested and Excluded (N=0)
Pneumonia (Infections and infestations) | 1 | 4 | 0 | NA
Unplanned intubation (Injury, poisoning and procedural complications) | 1 | 2 | 0 | NA — Assessed in the intraoperative or postoperative period of index hospitalization.
Aspiration pneumonitis/pneumonia (Infections and infestations) | 0 | 2 | 0 | NA
Pneumothorax with chest tube (Injury, poisoning and procedural complications) | 2 | 0 | 0 | NA
Stroke/cerebral vascular attack (Nervous system disorders) | 2 | 3 | 0 | NA
Transfusion of packed red blood cells (Injury, poisoning and procedural complications) | 7 | 5 | 0 | NA — Required high volume transfusion.
Intensive care unit admission (Injury, poisoning and procedural complications) | 2 | 5 | 0 | NA — Assessed during index hospitalization.
Death (General disorders) | 8 | 6 | 4 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | NA
Hypercalcemia/urinary tract infection (Infections and infestations) | 0 | 1 | 0 | NA
Myocardial infarction (Cardiac disorders) | 2 | 1 | 1 | NA
Deep incisional surgical site infection (Infections and infestations) | 0 | 2 | 0 | NA
Acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | NA
Hip dislocation (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | NA
Fall (Injury, poisoning and procedural complications) | 5 | 4 | 0 | NA
Surgical hardware removal (Injury, poisoning and procedural complications) | 1 | 1 | 0 | NA
Severe aortic stenosis (Cardiac disorders) | 0 | 1 | 0 | NA
Superficial incisional surgical site infection (Infections and infestations) | 1 | 1 | 0 | NA
Maxillary sinus tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA
Abdominal swelling (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Dysphagia/dysphonia (Gastrointestinal disorders) | 1 | 0 | 0 | NA
T12-L1 spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA
Ulcers (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | NA
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | NA
Eye surgery (Eye disorders) | 2 | 0 | 0 | NA
Cardiac arrest requiring cardiopulmonary resuscitation (Cardiac disorders) | 4 | 0 | 2 | NA
Bone fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | NA
Pituitary tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | NA — Surgical removal requiring hospitalization.
Avascular necrosis of femoral head (Injury, poisoning and procedural complications) | 1 | 1 | 0 | NA
Hypotension (General disorders) | 0 | 1 | 0 | NA
Inguinal hernia (Surgical and medical procedures) | 0 | 1 | 0 | NA
Total knee arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | NA
Non-ST-elevation myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | NA
Pelvic ring fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Cholecystitis/cholecystectomy (Surgical and medical procedures) | 0 | 1 | 0 | NA
Leg pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Carotid endarterectomy (Surgical and medical procedures) | 0 | 1 | 0 | NA
Respiratory distress (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Leg surgery (Surgical and medical procedures) | 1 | 0 | 1 | NA — Surgical repair of knee and foot requiring hospital readmission.
Knee replacement surgery (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Altered mental status (Psychiatric disorders) | 1 | 0 | 0 | NA
Tibia/fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | NA
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1 | 1 | NA
Chest pain (General disorders) | 1 | 0 | 0 | NA
Organ/space surgical site infection (Infections and infestations) | 1 | 1 | 0 | NA
Dysarthria (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | NA
Melena (Gastrointestinal disorders) | 1 | 0 | 0 | NA
Seizure (Nervous system disorders) | 1 | 0 | 0 | NA
Failed open reduction internal fixation of patella (Injury, poisoning and procedural complications) | 0 | 1 | 0 | NA
Liver failure (Endocrine disorders) | 0 | 0 | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: Usual General Anesthesia Care (N=56) | Experimental: Optimized General Anesthesia Care (N=53) | Mini Mental State Exam (N=22) | Tested and Excluded (N=0)
Superficial incisional surgical site infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 0
Transfusion of packed red blood cells (Injury, poisoning and procedural complications) | 21 | 17 | 0 | 0
Organ/space surgical site infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Limited availability of subjects meeting inclusion criteria resulting in early termination (lack of funding) before meeting target enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT02604459/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/59/NCT02604459/ICF_001.pdf